CLINICAL TRIAL: NCT00423943
Title: Modafinil for Treatment of Cognitive Dysfunction in Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Michael Minzenberg, MD, Principal Investigator, University of California, Davis
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 200513585-1
Record Dates: First submitted 2007-01-16; First posted 2007-01-18 (Estimated); Results first posted 2017-09-29 (Actual); Last update posted 2017-09-29 (Actual); Status verified 2017-08

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: cognition; memory
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- D (Experimental): modafinil
  Interventions: Drug: modafinil
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: modafinil — 200 milligrams daily dose
  Other Names: Provigil
  Arms: D
Drug: Placebos — capsule containing placebo
  Arms: Placebo

SUMMARY:
Patients with schizophrenia have problems in thinking, known as cognitive dysfunction. This appears to be responsible for their difficulties in social and occupational functioning. One particular cognitive function that may be important for schizophrenia is called context processing. This refers to the ability to properly use information in the environment to guide thinking and behavior so that it is appropriate to the present circumstance. Problems with this function may explain why patients with schizophrenia think and act in unusual ways, and often have problems managing aspects of their lives that healthy adults take for granted. This cognitive function depends on a region of the brain called the prefrontal cortex, which shows impaired function in schizophrenia as well. Unfortunately, the biochemical aspects of this dysfunction are presently unknown, and it is not clear whether current psychiatric medications can improve this function. A recent FDA-approved medication that may improve this function is modafinil. Studies in animals and healthy adults show that this medication can improve cognitive functions which are related to context processing. We plan to study the effects of modafinil on context processing and the brain activity that underlies this function. We will use functional MRI and electrophysiology to examine the effects of modafinil, both after a single dose and after sustained (4 week) treatment. We predict that when patients receive modafinil they will perform better on cognitive tests and have improved activity in the regions of the brain that are responsible for these cognitive processes.

DETAILED DESCRIPTION:
Schizophrenia is a disorder of cognition. The cognitive deficits of schizophrenia are present at the onset of the disorder, prior to medication exposure, are persistent during periods of remission, and are strongly related to functional outcome. These deficits prominently include prefrontal-dependent functions. While existing medications effectively treat psychotic symptoms, they exhibit modest benefit at best for cognitive dysfunction. Studies of cognition in animal models indicate that the neurotransmitter systems that mediate prefrontal-dependent cognitive processes are not generally augmented by existing antipsychotic medications. Therefore, advances in the treatment of schizophrenia will require the study of agents with novel pharmacological profiles to establish their potential to remediate cognitive dysfunction.

Advances in understanding the mechanism of action of these agents will also require the integration of pharmacology with a sophisticated methodology for testing cognition. This goal has been strongly pursued in recent years with the use of functional magnetic resonance imaging (fMRI) to study pharmacological effects on cognition. fMRI studies have identified the cortical network subserving cognitive control and working memory, which are consistently impaired among schizophrenia patients. The study of medication effects on these processes with fMRI (pharmaco-fMRI) will permit the more precise delineation of the cognitive mechanisms amenable to pharmacological intervention.

This study will use fMRI to study the effects of modafinil on the functional neuroanatomy underlying prefrontal cognitive processes. Modafinil is an FDA-approved medication with a unique pharmacological profile and an increasing range of off-label indications. Its neurochemical effects in animal models include elevation of extracellular dopamine (DA), noradrenaline (NA) and glutamate in the neocortex. This profile is favorable for the enhancement of prefrontal cognitive processes. These neurochemical effects also appear to be selective for cortical versus subcortical brain regions, suggesting that modafinil may have minimal effects on psychotic symptoms, or extrapyramidal, autonomic and hormonal side effects. In addition, it differs from amphetamine in structure, neurochemical profile and behavioral effects, with a lower risk of addictive or cerebrovascular effects. Recent studies in animal models, healthy adults and adults with psychiatric and neurological disorders indicate that modafinil improves prefrontal cognitive functions. This suggests that modafinil is a leading candidate for the treatment of cognitive dysfunction in schizophrenia. We aim to test modafinil effects on these processes in healthy adults, in order to evaluate modafinil effects on normal-range cognition, and then evaluate the remediation of deficits in these functions in individuals with schizophrenia, both in a single-dose trial and followed by a trial of sustained treatment.

Comparison 1. The effect in healthy adults and adults with schizophrenia/schizoaffective disorder, of Modafinil 200 milligrams single oral dose versus placebo (double-blind, balanced crossover design), on cognitive control task performance, and on activity of dorsolateral prefrontal cortical (DLPFC) during context processing, and anterior cingulate cortex (ACC) during conflict monitoring phases of the task, both measured by fMRI.

Comparison 2. The effect in adults with schizophrenia/schizoaffective disorder, of 4-week randomized, double-blind treatment with Modafinil 200 milligrams daily versus placebo, on cognitive control task performance, and on activity of dorsolateral prefrontal cortical (DLPFC) during context processing, and anterior cingulate cortex (ACC) during conflict monitoring phases of the task, both measured by fMRI.

ELIGIBILITY:
Inclusion Criteria:

* adults age 18-54
* diagnosis of schizophrenia or schizoaffective disorder, or healthy with no personal or family history of mental illness
* able to provide informed consent

Exclusion Criteria:

* history of significant head injury or other neurological illness
* active psychiatric illness requiring significant acute care
* significant intellectual impairment (e.g. standardized full-scale IQ < 70)
* history of medical illness or treatment that either interferes with experimental measures (e.g. cerebrovascular disease, anemias, etc.) or is associated with significant increase in risk from modafinil treatment (e.g. cardiac disease)
* significant active substance abuse
* presence of ferromagnetic foreign body or prosthesis
* active pregnancy
* active treatment with medications that have drug interactions with modafinil

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2005-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Minzenberg, MD, Principal Investigator — University of California, Los Angeles; Cameron S Carter, MD, Principal Investigator — University of California Davis School of Medicine
Locations (1):
- University of California Los Angeles School of Medicine, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Drug: modafinil
  modafinil: 200 milligrams daily dose
- Placebo: placebo
  modafinil: 200 milligrams daily dose
Period: Overall Study
Arm/Group | Drug | Placebo
Started | 19 | 14
Completed | 16 | 13
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Drug | Placebo | Total
Number analyzed (Participants) | 19 | 14 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 14 | 33
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.4 (7.7) | 25.8 (8.9) | 26.2 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 15 | 11 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 4
  Not Hispanic or Latino | 15 | 14 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 17 | 7 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 14 | 33

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Accuracy on High-control (i.e., Difficult) Condition of Preparing to Overcome Prepotency Task
Description: Accuracy change on high-control (i.e., difficult) condition of Preparing to Overcome Prepotency (POP) Task. For high-control condition (red-cue), subjects responded in the incongruent direction (eg, for a right-pointing arrow, press the left button, and vice versa). Increased values indicate improved performance.
Time Frame: Baseline, 4 weeks
Measure: Mean (Standard Deviation); unit: percent change in accuracy
Arm/Group | Drug | Placebo
Number analyzed (Participants) | 19 | 14
percent change in accuracy | 8.6 (9.8) | 9.2 (9.7)

2. Primary Outcome: Control-related BOLD Signal Change in Locus Coeruleus
Description: BOLD signal change on high-control (i.e. difficult) condition versus low-control (i.e. easy) condition, on Preparing to Overcome Prepotency Task, measured by fMRI after 4-week treatment.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: beta coefficient of BOLD signal change
Arm/Group | Drug | Placebo
Number analyzed (Participants) | 19 | 14
beta coefficient of BOLD signal change | -0.05 (0.63) | -0.74 (1.28)

3. Primary Outcome: Gamma Power Change in Count of Clusters
Description: Power in Gamma frequency range by scalp electrophysiology after single-dose and after 4-week treatment: Count of Clusters (defined as those with statistically-significant Task-Related Increase, i.e. relatively larger value of wavelet coefficient in wavelet analysis of signal) for high-control (i.e. difficult) condition versus Low-control (i.e. easy) condition, in Oscillatory Power in Time-Frequency Spectrogram. Increased values indicate improved function.
Time Frame: 4 weeks
Population: 2 subjects in the Drug arm refused to perform EEG.
Measure: Mean (Standard Deviation); unit: Count of Positive Power Clusters
Arm/Group | Drug | Placebo
Number analyzed (Participants) | 14 | 13
Count of Positive Power Clusters | 44 (12) | 17 (5)

4. Secondary Outcome: Change in Positive Symptoms
Description: Change in Average score (range 0-5) on the Scale for Assessment of Positive Symptoms (SAPS) from baseline to 4 week time-point, ranging from 0 (absent) to 5 (severe). Decreased values indicate improved clinical status (lesser symptom severity).
Time Frame: Baseline, 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drug | Placebo
Number analyzed (Participants) | 19 | 14
units on a scale | 0.80 (0.82) | 0.58 (0.56)

5. Secondary Outcome: Change in Negative Symptoms
Description: Change in average score, ranging from 0 (absent) to 5 (severe), on on Scale for the Assessment of Negative Symptoms (SANS) from baseline to 4-week time-point. Decreased values indicate improved clinical status (lesser symptom severity).
Time Frame: Baseline, 4 weeks
Measure: Mean (Standard Deviation); unit: units on SANS scale
Arm/Group | Drug | Placebo
Number analyzed (Participants) | 19 | 14
units on SANS scale | 1.88 (1.04) | 2.12 (1.15)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Drug | Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/14
Other Adverse Events (participants affected / at risk) | 0/19 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes